CLINICAL TRIAL: NCT02551861
Title: A Randomized, Open-Label Study of Daclatasvir and Sofosbuvir With or Without Ribavirin for 8 Weeks in Treatment-Naïve, Non-Cirrhotic Subjects Infected With Chronic HCV Genotype 3
Brief Title: A Randomized, Open-Label Study of Daclatasvir and Sofosbuvir With or Without Ribavirin for 8 Weeks in Treatment-Naïve, Non-cirrhotic Subjects Infected With Chronic Hepatitis C Virus (HCV) Genotype 3
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI444-377; 2015-003468-36 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daclatasvir + Sofosbuvir (Active Comparator): Daclatasvir 60mg tablet and Sofosbuvir 400mg tablet oral dosing once daily for 8 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir
- Daclatasvir + Sofosbuvir + Ribavirin (Active Comparator): Daclatasvir 60mg tablet + Sofosbuvir 400mg tablet+ Ribavirin 1000-1200mg tablet(weight based dosing) oral dosing split into am and pm once daily for 8 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Daclatasvir
Drug: Sofosbuvir
Drug: Ribavirin
  Arms: Daclatasvir + Sofosbuvir + Ribavirin

SUMMARY:
The purpose of this study is to determine if 8 weeks of Daclatasvir plus Sofosbuvir with or without Ribavirin is safe and effective in the treatment of genotype 3 hepatitis C infected patients without advanced fibrosis or liver cirrhosis who have never been treated previously.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Genotype 3
* HCV RNA < 2000000 IU/mL
* Never taken HCV medication
* Absence of advanced fibrosis or cirrhosis
* Body mass index (BMI) 18-40 kg/m^2

Exclusion Criteria:

* Infection with HCV other than genotype 3 (GT3); Mixed infections of any genotype
* Previously taken HCV medication
* Liver Cirrhosis
* Evidence of decompensated liver disease
* HIV/ hepatitis B virus (HBV) coinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with sustained virologic response (SVR12) treated with Daclatasvir + Sofosbuvir (DCV+SOF) | Post Treatment Follow up Week 12
  SVR12 defined as HCV RNA < LLOQ target detected (TD) or target not detected (TND) at follow-up Week 12 in subjects treated with 8 weeks of DCV+SOF therapy or DCV+SOF+RBV therapy

SECONDARY OUTCOMES:
Safety measured by number of incidence of deaths, serious adverse events (SAE)s, discontinuation due to adverse events (AE)s, Grade 3/4 AEs and Grade 3/4 laboratory abnormalities observed from clinical laboratory testing | Approximately 1.5 years
Antiviral activity measured by the proportion of subjects who achieve HCV RNA < lower limit of quantification (LLOQ) - at during and after treatment in each treatment arm | Post treatment follow up Week 24
Proportion of subjects with CC, CT or TT IL28B genotype who achieve SVR12 in each treatment arm | Post Treatment Follow up Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- Canada (5):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Toronto, Ontario
- France (6):
  - Local Institution, Créteil
  - Local Institution, Limoges
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Vandœuvre-lès-Nancy

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx